CLINICAL TRIAL: NCT04244773
Title: Substudy of Efficacy, Safety and Toxicology of Electronic Nicotine Delivery Systems as an Aid for Smoking Cessation (ESTxENDS Trial)- the Micronuclei Substudy of ESTxENDS
Brief Title: ESTxENDS Trial: MN Substudy - Micronuclei in Buccal Epithelium, a Surrogate Measure of Future Cancer Risk, Induced by Electronic Nicotine Delivery Systems (ENDS/Vaporizer/E-cig)
Acronym: ESTxENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Lausanne (Other); University of Geneva, Switzerland (Other); University of Zurich (Other); State Hospital, St. Gallen (Other Government); Swiss National Science Foundation (Other); Krebsforschung Schweiz, Bern, Switzerland (Other); Federal Office of Public Health, Switzerland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-02332i
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; Micronuclei
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Masking Description: Statisticians and laboratory personnel will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: ENDS and smoking cessation (Experimental)
  Interventions: Other: ENDS (vaporizer/e-cig) and smoking cessation counseling
- Control group: Smoking cessation counseling (Active Comparator)
  Interventions: Other: Smoking cessation counseling

INTERVENTIONS:
Other: ENDS (vaporizer/e-cig) and smoking cessation counseling — Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Intervention group: ENDS and smoking cessation
Other: Smoking cessation counseling — Participants in the control group will receive smoking cessation counseling only. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Control group: Smoking cessation counseling

SUMMARY:
--> This is a substudy of the main ESTxENDS trial (NCT03589989). Micronuclei in buccal epithelial outcomes should be considered secondary outcomes of the main smoking cessation outcome formulated in NCT03589989.

Cigarette smoking is the leading cause of preventable death in Switzerland and still more than a quarter of the Swiss population smokes cigarettes. Recently, electronic nicotine delivery systems (ENDS; also called vaporizer, e-cigarette or electronic cigarette) have become popular with smokers who want to stop smoking or reduce their exposure to inhaled chemicals since ENDS use appears to be safer than tobacco smoking.

The micronucleus cytologic assay test was originally developed to screen for drug toxicity in bone marrow samples from mammals. The technique identifies micronuclei on smears obtained by oral cavity exfoliation and indicate genomic instability. Buccal MNs may predict cancer risk for the upper aerodigestive tract. The HUman MicroNucleus project on eXfoLiated buccal cells (HUMNXL) found MN counts gradually increased during the progression from normal mucosal to precancerous lesions to carcinoma. MN assessment discriminates between exposure to tobacco smoke in smokers and in non-smokers, and has been tested on a small number of ENDS users.

For the main ESTxENDS trial (NCT03589989), cigarette smokers motivated to quit smoking cigarettes will be included. Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants in the control group will receive smoking cessation counseling only. All participants will be followed over a 24-month period. Measures of MN frequency will test the potential effect of ENDS use on cancer-related outcomes, in particular incident of mouth-, lung- and kidney- cancers.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Persons aged 18 or older
* Currently smoking 5 or more cigarettes a day for at least 12 months
* Willing to try to quit smoking within the next 3 months,
* Persons providing a valid phone number, a valid email address and/or a valid postal address.

Exclusion Criteria:

Known hypersensitivity or allergy to contents of the e-liquid Participation in another study with investigational drug within the 30 days preceding the baseline visit and during the present study where interactions are to be expected

* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the scheduled study intervention, i.e. within the first 6-months of the study
* Persons having used ENDS regularly in the 3 months preceding the baseline visit
* Persons having used nicotine replacement therapy (NRT) or other medications with demonstrated efficacy as an aid for smoking cessation such as varenicline or bupropion within the 3 months preceding the baseline visit
* Persons who cannot attend the 6- month follow-up visit for any reason
* Cannot understand instructions delivered in person or by phone, or otherwise unable to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Frequency of buccal micronuclei_1 | Baseline
  MN frequency will be calculated as number of cells that contain MNs divided by the total number counted. A minimum of 1000 cells will be counted per participant.
Frequency of buccal micronuclei_2 | 6 months post quit date
  MN frequency will be calculated as number of cells that contain MNs divided by the total number counted. A minimum of 1000 cells will be counted per participant.
Frequency of buccal micronuclei_3 | 12 months post quit date
  MN frequency will be calculated as number of cells that contain MNs divided by the total number counted. A minimum of 1000 cells will be counted per participant.
Frequency of buccal micronuclei_4 | 24 months post quit date
  MN frequency will be calculated as number of cells that contain MNs divided by the total number counted. A minimum of 1000 cells will be counted per participant.

SECONDARY OUTCOMES:
Change of frequency of buccal micronuclei | Change from baseline to 6,12, 24 months post quit date
  MN frequency will be calculated as number of cells that contain MNs divided by the total number counted. A minimum of 1000 cells will be counted per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, Prof.Dr.med., Study Director — Berner Institut für Hausarztmedizin; Universität Bern; Nancy Hopf, PD Dr., Principal Investigator — Centre universitaire de médecine générale et santé publique, Lausanne
Locations (5):
- Switzerland (5):
  - Unisanté, Centre universitaire de médecine générale et santé publique, Université de Lausanne, Lausanne, Canton of Vaud
  - University Clinic for General Internal Medicine, Bern University Hospital, Bern
  - Département de médecine interne, Hôpitaux universitaires de Genève, Geneva
  - Lungenzentrum, Klinik für Pneumologie und Schlafmedizin, Kantonsspital St. Gallen, Sankt Gallen
  - Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich, Zurich

REFERENCES:
- [Background] Bloching M, Hofmann A, Lautenschlager C, Berghaus A, Grummt T. Exfoliative cytology of normal buccal mucosa to predict the relative risk of cancer in the upper aerodigestive tract using the MN-assay. Oral Oncol. 2000 Nov;36(6):550-5. doi: 10.1016/s1368-8375(00)00051-8. PMID 11036250
- [Background] Casartelli G, Bonatti S, De Ferrari M, Scala M, Mereu P, Margarino G, Abbondandolo A. Micronucleus frequencies in exfoliated buccal cells in normal mucosa, precancerous lesions and squamous cell carcinoma. Anal Quant Cytol Histol. 2000 Dec;22(6):486-92. PMID 11147304
- [Background] Franco T, Trapasso S, Puzzo L, Allegra E. Electronic Cigarette: Role in the Primary Prevention of Oral Cavity Cancer. Clin Med Insights Ear Nose Throat. 2016 Oct 17;9:7-12. doi: 10.4137/CMENT.S40364. eCollection 2016. PMID 27773997
- [Background] Nersesyan A, Muradyan R, Kundi M, Knasmueller S. Impact of smoking on the frequencies of micronuclei and other nuclear abnormalities in exfoliated oral cells: a comparative study with different cigarette types. Mutagenesis. 2011 Mar;26(2):295-301. doi: 10.1093/mutage/geq092. Epub 2010 Nov 2. PMID 21044989
- [Background] El-Setouhy M, Loffredo CA, Radwan G, Abdel Rahman R, Mahfouz E, Israel E, Mohamed MK, Ayyad SB. Genotoxic effects of waterpipe smoking on the buccal mucosa cells. Mutat Res. 2008 Aug-Sep;655(1-2):36-40. doi: 10.1016/j.mrgentox.2008.06.014. PMID 18662802
- [Background] Tolbert PE, Shy CM, Allen JW. Micronuclei and other nuclear anomalies in buccal smears: a field test in snuff users. Am J Epidemiol. 1991 Oct 15;134(8):840-50. doi: 10.1093/oxfordjournals.aje.a116159. PMID 1951279